CLINICAL TRIAL: NCT05274815
Title: A Multicentre, Single-arm, Phase 3b Efficacy and Safety Study of Tezepelumab 210 mg Administered Subcutaneously to Reduce Oral Corticosteroid Use in Adult Participants With Severe Asthma on High-dose Inhaled Corticosteroid Plus Long-acting β2 Agonist and Long-term Oral Corticosteroid Therapy (WAYFINDER)
Brief Title: Study to Evaluate Efficacy and Safety of Tezepelumab in Reducing Oral Corticosteroid Use in Adult Patients With Severe Asthma
Acronym: WAYFINDER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5180C00037; 2021-005457-85 (EudraCT Number)
Record Dates: First submitted 2022-01-27; First posted 2022-03-10 (Actual); Results first posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Asthma
Keywords: Asthma; Severe Asthma; Oral Corticosteroids
MeSH Terms: conditions — Asthma | interventions — tezepelumab

STUDY DESIGN:
Intervention Model Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tezepelumab (Experimental): Tezepelumab subcutaneous injection
  Interventions: Biological: Tezepelumab

INTERVENTIONS:
Biological: Tezepelumab — Tezepelumab subcutaneous injection

SUMMARY:
This is a study designed to evaluate efficacy and safety of Tezepelumab in reducing oral corticosteroid use in adult patients with severe asthma who are receiving oral corticosteroids with or without additional asthma controller medications.

DETAILED DESCRIPTION:
This is a multicentre, single-arm, phase 3b study designed to evaluate efficacy and safety of reducing daily oral corticosteroid use after initiation of 210 mg dose of Tezepelumab administered subcutaneously in patients with severe asthma receiving high-dose inhaled corticosteroid plus long-acting β2 agonist and oral corticosteroids with or without additional asthma controller medications.

ELIGIBILITY:
Main inclusion criteria:

* Age 18-80 years.
* Documented physician diagnosed asthma requiring continuous treatment with high-dose ICS plus a LABA for at least 6 months prior to Visit 1. The ICS and LABA can be contained within a combination product or given by separate inhalers.
* Documented long-term OCS therapy for asthma, equivalent to a daily dose of at least 5 mg and up to 40 mg of prednisone/prednisolone for at least 3 continuous months directly preceding Visit 1.
* Participant should be on a stable maintenance OCS dose for at least 4 weeks prior to Visit 1.
* Documented history of at least 1 asthma exacerbation event within 12 months prior to Visit 1.

Other inclusion criteria per protocol apply.

Main exclusion criteria:

* Pulmonary disease or systemic diseases, other than asthma associated with elevated peripheral EOS counts.
* Any disorder or major physical impairment that is not stable and could affect the safety of the participant throughout the study, influence the findings of the study or the interpretation, or impede the participant's ability to complete the entire duration of study.
* History of cancer.
* History of a clinically significant infection requiring treatment with antibiotics, antiviral or additional corticosteroid medications finalised < 2 weeks before Visit 1.
* A helminth parasitic infection diagnosed within 6 months prior to Visit 1 that has not been treated with, or has failed to respond to, standard of care therapy.
* Current smokers or participants with smoking history ≥ 10 pack-years and participants using vaping products, including electronic cigarettes.
* History of chronic alcohol or drug abuse within 12 months prior to Visit 1.
* Tuberculosis requiring treatment within the 12 months prior to Visit 1.
* History of known immunodeficiency disorder including a positive HIV test at Visit 1.
* Major surgery within 8 weeks prior to Visit 1 or planned surgical procedures requiring general anaesthesia or inpatient status for > 1 day during the conduct of the study.
* Coexistent inflammatory conditions for which long-term OCS doses are part of their maintenance treatment.
* Receipt of any marketed or investigational biologic agent within 4 months or 5 half-lives (whichever is longer) prior to Visit 1 or receipt of any investigational nonbiologic agent within 30 days or 5 half-lives (whichever is longest) prior to Visit 1. Participants enrolled in current or previous tezepelumab studies will not be included.
* Concurrent enrolment in another clinical study involving an IP.
* Treatment with systemic immunosuppressive/immunomodulating drugs, except for OCS used in the treatment of asthma/asthma exacerbations, within the last 12 weeks or 5 half-lives (whichever is longer) prior to Visit 1.
* History of anaphylaxis or documented immune complex disease (Type III hypersensitivity reactions) following any biologic therapy.
* Positive hepatitis B surface antigen, or hepatitis C virus antibody serology at screening, or a positive medical history for hepatitis B or C.
* Pregnant, breastfeeding, or lactating women.

Other exclusion criteria per protocol apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2024-09-09 (Actual); Study Completion 2024-09-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (67):
- United States (7):
  - Research Site, Newport Beach, California
  - Research Site, Newark, Delaware
  - Research Site, Loxahatchee Groves, Florida
  - Research Site, Ann Arbor, Michigan
  - Research Site, Toms River, New Jersey
  - Research Site, The Bronx, New York
  - Research Site, DuBois, Pennsylvania
- Argentina (11):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Mendoza
  - Research Site, Monte Grande
  - Research Site, Pilar
  - Research Site, Quilmes
  - Research Site, Ranelagh
  - Research Site, Rosario
  - Research Site, San Fernando
  - Research Site, San Juan Bautista
  - Research Site, San Miguel de Tucumán
- Belgium (4):
  - Research Site, Brussels (Woluwé-St-Lambert)
  - Research Site, Erpent
  - Research Site, Ghent
  - Research Site, Liège
- Bulgaria (4):
  - Research Site, Haskovo
  - Research Site, Razgrad
  - Research Site, Sofia
  - Research Site, Velika Tarnovo
- France (8):
  - Research Site, Antony
  - Research Site, Bordeaux
  - Research Site, Brest
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Nantes
  - Research Site, Nice
- Germany (5):
  - Research Site, Berlin
  - Research Site, Darmstadt
  - Research Site, Fürstenwalde
  - Research Site, Mainz
  - Research Site, Reinfeld (Holstein)
- Latvia (4):
  - Research Site, Daugavpils
  - Research Site, Jūrmala
  - Research Site, Riga
  - Research Site, Valmiera
- Mexico (3):
  - Research Site, Chihuahua City
  - Research Site, Guadalajara
  - Research Site, Monterrey
- Poland (8):
  - Research Site, Bychawa
  - Research Site, Chmielnik
  - Research Site, Gdansk
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Ostrowiec Świętokrzyski
  - Research Site, Sosnowiec
  - Research Site, Wroclaw
- Spain (7):
  - Research Site, Badalona
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Oviedo
  - Research Site, Santa Cruz de Tenerife
  - Research Site, Santander
  - Research Site, Seville
- United Kingdom (6):
  - Research Site, Belfast
  - Research Site, Bradford
  - Research Site, LE3 9QP
  - Research Site, London
  - Research Site, Nottingham
  - Research Site, Portsmouth

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of the timelines, please rerefer to the disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Jackson DJ, Lugogo NL, Gurnell M, Heaney LG, Korn S, Brusselle G, Chanez P, Del Olmo R, Llanos JP, Keeling N, Salapa K, Cook B, Parulekar AD, Kostikas K, Fogel R, Martin N, Chandarana SN. Oral corticosteroid reduction and discontinuation in adults with corticosteroid-dependent, severe, uncontrolled asthma treated with tezepelumab (WAYFINDER): a multicentre, single-arm, phase 3b trial. Lancet Respir Med. 2025 Nov 26:S2213-2600(25)00359-5. doi: 10.1016/S2213-2600(25)00359-5. Online ahead of print. PMID 41317738
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5180C00037&attachmentIdentifier=34d82b3c-095c-46d3-988d-684d6a36c498&fileName=D5180C00037_CSP_Redacted.pdf&versionIdentifier=
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5180C00037&attachmentIdentifier=c0811001-71fd-4900-8ccb-2c061b7cf697&fileName=D5180C00037_CSR_Synopsis.pdf&versionIdentifier=
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5180C00037&attachmentIdentifier=0ed21781-6d75-4e43-b87d-e42dfdc3186a&fileName=D5180C00037_SAP_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 305 participants were enrolled from 68 study sites across 11 countries, including sites in Argentina, Belgium, Bulgaria, France, Germany, Latvia, Mexico, Poland, Spain, UK, and USA.
Pre-assignment Details: Of the 305 participants that initiated treatment with tezepelumab, 7 were excluded from the efficacy and safety summary due to potential data fraud. Therefore, only 298 participants were included in the summaries.
Groups:
- Tezepelumab: Tezepelumab 210 mg was administered subcutaneously (SC) every 4 weeks (Q4W) for a total of 13 doses
  Induction phase (Week 0 to 4): At the screening visit, participants continued or were switched to prednisone or prednisolone. Participants started to receive tezepelumab treatment at Visit 2/Week 0 (baseline) and had to remain stable on their baseline oral corticosteroid (OCS) dose during this phase.
  OCS reduction and maintenance phase (Week 4 to Week 52): Initial OCS tapering was guided by an algorithm based on baseline OCS dose until the lowest stable OCS dose (OCS discontinued or no further OCS reduction possible) was reached or until Week 48; dosages were reduced in 2.5- to 5-mg increments weekly, every 2 weeks, or Q4W.
Period: Overall Study
Arm/Group | Tezepelumab
Started | 298
Completed | 273
Not Completed | 25
Not completed — Adverse Event | 1
Not completed — Death | 2
Not completed — Lost to Follow-up | 4
Not completed — Withdrawn from study due to investigator's decision | 1
Not completed — Withdrawn from study due to participant's decision to withdraw | 1
Not completed — Withdrawn from study due to severe non-compliance with the protocol | 1
Not completed — Withdrawn from study due to subject decision | 1
Not completed — Withdrawn due to participant's decision not to continue for personal and family reasons | 1
Not completed — Withdrawn from study due to the participant stopped visit; agreed to a telephone contact at Week 52 | 1
Not completed — Withdrawn from study due to randomization into closed cohort by mistake | 1
Not completed — Withdrawal by Subject | 11

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: included all enrolled participants who received at least one dose of tezepelumab, irrespective of their protocol adherence and continued participation in the study.
Groups:
- Tezepelumab: Tezepelumab 210 mg was administered SC Q4W for a total of 13 doses.
  Induction phase (Week 0 to 4): Participants received tezepelumab treatment at Visit 2/Week 0 (baseline) and had to remain stable on their baseline OCS dose during this phase.
  OCS reduction and maintenance phase (Week 4 to 52): Initial OCS tapering was guided by an algorithm based on baseline OCS dose until the lowest stable OCS dose (OCS discontinued or no further OCS reduction possible) was reached or until Week 48; dosages were reduced in 2.5- to 5-mg increments weekly, every 2 weeks, or Q4W OCS dose.
Arm/Group | Tezepelumab
Number analyzed (Participants) | 298
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at Screening Population: Full Analysis Set
  Years | 54.4 (12.0)
Age, Customized [Number; unit: Participants] — Age at Screening Population: Full Analysis Set
  Participants
    >=18 to <65 years | 231
    >=65 years | 67
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Full Analysis Set
  Participants
    Female | 206
    Male | 92
Race/Ethnicity, Customized [Number; unit: Participants] — Population: Full Analysis Set
  Participants
    Hispanic or Latino | 123
    Not Hispanic or Latino | 157
    Missing | 18
Race/Ethnicity, Customized [Number; unit: Participants] — Population: Full Analysis Set
  Participants
    Black or African American | 2
    American Indian or Alaska Native | 5
    White | 258
    Other | 15
    Not reported | 18
Region of Enrollment [Number; unit: Participants] — Full Analysis Set
  Participants
    Argentina | 80
    Belgium | 13
    Bulgaria | 36
    France | 18
    Germany | 22
    Latvia | 16
    Mexico | 41
    Poland | 40
    Spain | 8
    United States | 12
    United Kingdom | 12

OUTCOME MEASURES:

1. Primary Outcome: Proportion of the Participants Who Discontinued OCS Without Loss of Asthma Control at Week 28 and Week 52
Description: The proportion (expressed as a percentage) of participants who discontinued OCS without loss of asthma control is presented.
  Loss of asthma control was defined as asthma worsening or exacerbation. Asthma worsening was defined by an increase of Asthma Control Questionnaire 6 (ACQ-6) score ≥0.5 from baseline. Asthma exacerbation was defined by worsening of asthma symptoms that led to temporary bolus/burst of systemic corticosteroids (SCS; or a temporary increase in stable OCS background dose) for at least 3 consecutive days (a single depo-injectable dose of corticosteroids being considered equivalent to a 3-day bolus/burst of SCS), and/or an emergency room (ER) or urgent care visit requiring SCS, and/or inpatient hospitalisation, both due to asthma.
Time Frame: Week 28 and Week 52
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tezepelumab
Number analyzed (Participants) | 298
Percentage of participants
  Week 28 | 32.2 [26.9 to 37.8]
  Week 52 | 50.3 [44.5 to 56.2]

2. Primary Outcome: Proportion of the Participants Who Reduced Daily Prescribed Maintenance OCS Dose to ≤5 mg/Day Without Loss of Asthma Control at Week 28 and Week 52
Description: The proportion (expressed as a percentage) of the participants who reduced daily prescribed maintenance OCS dose to ≤5 mg/day without loss of asthma control at Week 28 and Week 52 is presented.
Time Frame: Week 28 and Week 52
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tezepelumab
Number analyzed (Participants) | 298
Percentage of participants
  Week 28 | 88.9 [84.8 to 92.3]
  Week 52 | 89.9 [85.9 to 93.1]

3. Secondary Outcome: Annual Asthma Exacerbation Rate (AAER) Over Week 28 and Over Week 52
Description: The AAER over Week 28 and over Week 52 is presented. The AAER was calculated as the total number of asthma exacerbations over the period (Week 28/52) divided by the total time at risk for the period (Week 28 or Week 52).
Time Frame: Week 28 and Week 52
Population: as for baseline characteristics
Measure: Number; unit: exacerbations/year
Arm/Group | Tezepelumab
Number analyzed (Participants) | 298
exacerbations/year
  Week 28 | 0.66
  Week 52 | 0.57

4. Secondary Outcome: Rate of Asthma Exacerbation Associated With Hospitalisation or ER Visit Over 28 Weeks and Over 52 Weeks
Description: The AAER for exacerbations associated with hospitalisation or ER visit over 28 weeks and over 52 weeks is presented. The AAER was calculated as the total number of asthma exacerbations over the period (Week 28/52) divided by the total time at risk for the period (Week 28 or Week 52).
Time Frame: Week 28 and Week 52
Population: as for baseline characteristics
Measure: Number; unit: exacerbations/year
Arm/Group | Tezepelumab
Number analyzed (Participants) | 298
exacerbations/year
  Week 28 | 0.13
  Week 52 | 0.11

5. Secondary Outcome: Rate of Asthma Exacerbation Associated With Hospitalisation Over 28 Weeks and Over 52 Weeks
Description: The AAER for exacerbations associated with hospitalisation over 28 weeks and over 52 weeks are presented. The AAER was calculated as the total number of asthma exacerbations over the period (Week 28/52) divided by the total time at risk for the period (Week 28 or Week 52).
Time Frame: Week 28 and Week 52
Population: as for baseline characteristics
Measure: Number; unit: exacerbations/year
Arm/Group | Tezepelumab
Number analyzed (Participants) | 298
exacerbations/year
  Week 28 | 0.06
  Week 52 | 0.05

6. Secondary Outcome: Proportion of the Participants Who Did Not Experience an Exacerbation Over 28 Weeks and Over 52 Weeks
Description: The proportion (expressed as a percentage) of participants who completed 28 or 52 weeks of treatment and did not experience an exacerbation over 28 weeks and over 52 weeks is presented.
Time Frame: Week 28 and Week 52
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tezepelumab
Number analyzed (Participants) | 298
Percentage of participants
  Week 28: number analyzed (Participants) | 288
  Week 28 | 76.0 [70.68 to 80.85]
  Week 52: number analyzed (Participants) | 275
  Week 52 | 66.9 [61.01 to 72.44]

7. Secondary Outcome: Proportion of the Participants Who Did Not Experience an Exacerbation Associated With Hospitalisation or ER Visit Over 28 Weeks and Over 52 Weeks
Description: The proportion (expressed as a percentage) of participants who completed 28 or 52 weeks of treatment and did not experience an exacerbation associated with hospitalisation or ER visit over 28 weeks and over 52 weeks is presented.
Time Frame: Week 28 and Week 52
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tezepelumab
Number analyzed (Participants) | 298
Percentage of participants
  Week 28: number analyzed (Participants) | 288
  Week 28 | 95.5 [92.40 to 97.57]
  Week 52: number analyzed (Participants) | 275
  Week 52 | 92.7 [88.99 to 95.50]

8. Secondary Outcome: Proportion of the Participants Who Did Not Experience an Exacerbation Associated With Hospitalisation Over 28 Weeks and Over 52 Weeks
Description: The proportion (expressed as a percentage) of participants who completed 28 or 52 weeks of treatment and did not experience an exacerbation associated with hospitalisation over 28 weeks and over 52 weeks is presented.
Time Frame: Week 28 and Week 52
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Tezepelumab
Number analyzed (Participants) | 298
Percentage
  Week 28: number analyzed (Participants) | 288
  Week 28 | 97.9 [95.52 to 99.23]
  Week 52: number analyzed (Participants) | 275
  Week 52 | 96.0 [92.96 to 97.99]

9. Secondary Outcome: Proportion of the Participants With ≥50% Reduction From Baseline in Daily Maintenance OCS Dose at Week 28 and Week 52
Description: The proportion (expressed as a percentage) of participants with ≥50% reduction from baseline in daily maintenance OCS dose at Week 28 and Week 52 is presented.
  The baseline OCS dose is the prescribed OCS dose prior to first dose of investigational product (IP). The final daily OCS dose was defined as the last dose reported by participants with asthma stability verified (no change in OCS dose for at least 2 consecutive weeks).
Time Frame: Week 28 and Week 52
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tezepelumab
Number analyzed (Participants) | 298
Percentage of participants
  Week 28 | 76.8 [71.6 to 81.5]
  Week 52 | 81.9 [77.0 to 86.1]

10. Secondary Outcome: Categorised Percent Reduction From Baseline in the Daily Maintenance OCS Dose at Week 28 and Week 52
Description: The categorised percent reduction from baseline in the daily maintenance OCS dose (categories: ≥90% to ≤100% reduction, ≥75% to <90% reduction, ≥50% to <75% reduction, >0% to <50% reduction, no change or any increase) at Week 28 and Week 52 is presented.
  The baseline OCS dose is the prescribed OCS dose prior to first dose of IP. The final daily OCS dose was defined as the last dose reported by participants with asthma stability verified (no change in OCS dose for at least 2 consecutive weeks).
Time Frame: Week 28 and Week 52
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Tezepelumab (Week 28): Participants with OCS-dependent asthma with high-dose ICS plus LABA with or without additional asthma controller and with at least 1 asthma exacerbation in the prior year who received at least one dose of tezepelumab
Arm/Group | Tezepelumab (Week 28)
Number analyzed (Participants) | 298
Percentage of participants
  Week 28: ≥90% to ≤100% reduction | 35.2 [29.8 to 41.0]
  Week 28: ≥75% to <90% reduction | 14.1 [10.4 to 18.6]
  Week 28: ≥50% to <75% reduction | 27.5 [22.5 to 33.0]
  Week 28: >0% to <50% reduction | 8.1 [5.2 to 11.7]
  Week 28: No change or any increase | 15.1 [11.2 to 19.7]
  Week 52: ≥90% to ≤100% reduction | 52.0 [46.2 to 57.8]
  Week 52: ≥75% to <90% reduction | 9.1 [6.1 to 12.9]
  Week 52: ≥50% to <75% reduction | 20.8 [16.3 to 25.9]
  Week 52: >0% to <50% reduction | 4.0 [2.1 to 6.9]
  Week 52: No change or any increase | 14.1 [10.4 to 18.6]

11. Secondary Outcome: Absolute Change From Baseline in Daily Maintenance OCS Dose at Week 28 and Week 52
Description: The absolute change from baseline in daily maintenance OCS dose at Week 28 and Week 52 is presented.
  The baseline OCS dose is the prescribed OCS dose prior to first dose of IP. The final daily OCS dose was defined as the last dose reported by participants with asthma stability verified (no change in OCS dose for at least 2 consecutive weeks).
Time Frame: Week 28 and Week 52
Population: The analysis was done on the Full Analysis Set, including only subjects with an OCS dose at baseline and at least one non-missing post baseline value.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Tezepelumab
Number analyzed (Participants) | 298
mg
  Week 28 | -6.951 (5.596)
  Week 52 | -7.704 (6.294)

12. Secondary Outcome: Percent Change From Baseline in Daily Maintenance OCS Dose at Week 28 and Week 52
Description: The percent change from baseline in daily maintenance OCS dose at Week 28 and Week 52 is presented.
  The baseline OCS dose is the prescribed OCS dose prior to first dose of IP. The final daily OCS dose was defined as the last dose reported by participants with asthma stability verified (no change in OCS dose for at least 2 consecutive weeks).
Time Frame: Week 28 and Week 52
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Tezepelumab
Number analyzed (Participants) | 298
Percentage change
  Week 28 | -61.919 (41.773)
  Week 52 | -69.844 (43.666)

13. Secondary Outcome: Change From Baseline in Post-bronchodilator FEV1 at Week 28 and Week 52
Description: The change from baseline in post-bronchodilator FEV1 at Week 28 and Week 52 is presented. Baseline was defined as the last measurement at or prior first dose of IP.
  FEV1 = forced expiratory volume in 1 second
Time Frame: Week 28 and Week 52
Population: The analysis was done on the FAS, including only subjects with post-BD FEV1 at baseline and at least one non-missing post baseline value.
Measure: Mean (Standard Deviation); unit: liter (L)
Arm/Group | Tezepelumab
Number analyzed (Participants) | 298
liter (L)
  Week 28: number analyzed (Participants) | 242
  Week 28 | 0.0885 (0.3405)
  Week 52: number analyzed (Participants) | 232
  Week 52 | 0.0737 (0.3559)

14. Secondary Outcome: Change From Baseline in ACQ-6 at Week 28 and Week 52
Description: The Asthma Control Questionnaire 6 (ACQ-6) is a 6-item questionnaire which includes the following questions: 1) Awakening at night by symptoms, 2) Limitations of normal daily activities, 3) Waking in the morning with symptoms, 4) Dyspnoea, 5) Wheeze, and 6) Daily rescue medication. Questions were scored from 0 (totally controlled) to 6 (severely uncontrolled) and the ACQ-6 score was computed as the unweighted mean of the responses to the 6 questions. Higher scores indicate poorer outcomes.
  The change from baseline in ACQ-6 at Week 28 and Week 52 is presented.
Time Frame: Week 28 and Week 52
Population: The analysis is done on the FAS, including only subjects with ACQ-6 score at baseline and at least one non-missing post baseline value.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Tezepelumab
Number analyzed (Participants) | 298
Score on a scale
  Week 28: number analyzed (Participants) | 238
  Week 28 | -1.12 (1.00)
  Week 52: number analyzed (Participants) | 222
  Week 52 | -1.20 (1.09)

15. Secondary Outcome: Change From Baseline in Standardised AQLQ(s)+12 Total Score at Week 28 and Week 52
Description: The Asthma Quality of Life Questionnaire for 12 Years and Older (AQLQ[S]+12) is a questionnaire that measures the health-related quality of life experienced by asthma participants. Questions were scored from 7 (no impairment) to 1 (severe impairment). The overall score is calculated as the mean response to all questions. Higher scores indicate better outcomes.
  The change from baseline in standardised AQLQ(S)+12 total score at Week 28 and Week 52 is presented.
Time Frame: Week 28 and Week 52
Population: The analysis is done on the FAS, including only subjects with AQLQ(S)+12 total score at baseline and at least one non-missing post baseline value.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Tezepelumab
Number analyzed (Participants) | 298
Score on a scale
  Week 28: number analyzed (Participants) | 220
  Week 28 | 1.1455 (1.0419)
  Week 52: number analyzed (Participants) | 230
  Week 52 | 1.1932 (1.1551)

16. Secondary Outcome: Change From Baseline in SGRQ Total Score at Week 28 and Week 52
Description: The St. George's Respiratory Questionnaire (SGRQ) is a 50-item instrument developed to measure the health status of participants with airway obstruction diseases. The total score indicates the impact of disease on overall health status. The total score ranges for the SGRQ are 0-100, with higher scores indicating worse health status.
  The change from baseline in SGRQ total score at Week 28 and Week 52 is presented.
Time Frame: Week 28 and Week 52
Population: The analysis is done on the FAS, including only subjects with SGRQ total score at baseline and at least one non-missing post baseline value.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Tezepelumab
Number analyzed (Participants) | 298
score
  Week 28: number analyzed (Participants) | 216
  Week 28 | -16.2919 (18.1489)
  Week 52: number analyzed (Participants) | 226
  Week 52 | -16.6593 (18.7749)

ADVERSE EVENTS:
Time Frame: From the date of first dose of IP until study completion or withdrawal date, up to 64 weeks
Description: Only events that fall into the following categories were collected in this study: serious AEs, AEs leading to discontinuation of IP, and AEs of special interest. Participants with multiple occurrences in the same category were counted once per category regardless of the number of occurrences.
Arm/Group | Tezepelumab
All-Cause Mortality (participants affected / at risk) | 2/298
Serious Adverse Events (participants affected / at risk) | 28/298
Other Adverse Events (participants affected / at risk) | 4/298
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tezepelumab (N=298)
Adrenocortical insufficiency acute (Endocrine disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1)
Bronchitis bacterial (Infections and infestations) | 1 (1)
Angina pectoris (Cardiac disorders) | 2 (2)
Covid-19 (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 13 (15)
Aortic valve incompetence (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (3)
Cardiac failure (Cardiac disorders) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1)
Tachycardia foetal (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tezepelumab (N=298)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator shall be entitled to publish the results of, or make presentations related to, the Study, provided that any publications or presentations to be made within 2 years after completion of the Study shall require the Sponsor's prior written consent.

DOCUMENTS (2):
  • Study Protocol (2022-11-10): https://cdn.clinicaltrials.gov/large-docs/15/NCT05274815/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-09): https://cdn.clinicaltrials.gov/large-docs/15/NCT05274815/SAP_001.pdf